CLINICAL TRIAL: NCT01952132
Title: Phase 2 Randomized, Double-blind, Placebo-controlled, Sequential Dose Escalation Cohort Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of OMS643762 in Psychiatrically Stable Schizophrenia Subjects
Brief Title: Safety, Tolerability, and Pharmacokinetics of OMS643762 in Psychiatrically Stable Schizophrenia Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS824-SCZ-001
Record Dates: First submitted 2013-09-19; First posted 2013-09-27 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- OMS643762 Low Dose (Experimental): Orally administering OMS643762 low dose daily for 14 days
  Interventions: Drug: OMS643762
- OMS643762 High Dose (Experimental): Orally administering OMS643762 high dose daily for 14 days
  Interventions: Drug: OMS643762
- Placebo (Placebo Comparator): Orally administering placebo daily for 14 days
  Interventions: Drug: Placebo
- OMS643762 Medium Dose (Experimental): Orally administering OMS643762 medium dose daily for 14 days
  Interventions: Drug: OMS643762

INTERVENTIONS:
Drug: OMS643762
  Other Names: OMS824
  Arms: OMS643762 High Dose; OMS643762 Low Dose; OMS643762 Medium Dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability and pharmacokinetics of OMS643762 (the study drug) in psychiatrically stable schizophrenia patients.

ELIGIBILITY:
Inclusion Criteria:

* Competent to provide informed consent.
* Voluntarily provide informed consent and Health Insurance Portability and Accounting Act (HIPAA) Authorization in accordance with local regulations and governing Institutional Review Board (IRB) requirements prior to any procedures or evaluations performed specifically for the sole purpose of the study.
* Have a diagnosis of schizophrenia as defined in DSM-IV-TR.
* Are from 18 to 55 years of age inclusive at the screening visit.
* Have stable schizophrenia symptomatology for greater than or equal to three months at the screening visit, in the opinion of the investigator.
* For enrollment to Cohorts 1 and 2, have not taken any oral antipsychotic medication for at least seven days or any parenteral antipsychotic medication for at least 30 days prior to randomization. Subjects should have been on a stable medication regimen for greater than or equal to two months at the screening visit.
* For enrollment to Cohorts 3, 4, and 5, have been on a stable medication regimen for greater than or equal to two months at the screening visit.
* Have normal clinical laboratory test results and ECG, or results with minor deviations, which are not considered to be clinically significant by the investigator.
* If able to reproduce, agree to use an acceptable method of birth control (e.g., condom and spermicide, oral birth control which has been stable for 30 days) or agree to remain abstinent from Visit 2 until 90 days after the last dose of study drug for males and 30 days after the last dose of study drug for females.

Exclusion Criteria:

* Have a history of lactose intolerance or allergy to dairy products.
* Are pregnant or lactating.
* Have a history or presence of significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorders which, in the opinion of the investigator, increases the risk of the study drug or may confound the interpretation of study measures.
* Have a history of alcohol dependence (within 12 months of screening) or abuse (within six months of screening) as defined by DSM-IV-TR or consume excessive amounts of alcohol, in the opinion of the investigator.
* Have a history of substance dependence (within 12 months of screening) or abuse (within six months of screening) as defined by DSM-IV-TR (with the exception of nicotine and caffeine). Positive results on drug screening will be exclusionary unless the patient has a valid prescription for the medication (i.e., benzodiazepines).
* Have unstable depression, in the opinion of the investigator.
* Have experienced EPS within 30 days prior to Visit 1.
* Are currently taking clozapine.
* Are currently taking aripiprazole (for enrollment to Cohorts 1 and 2).
* Have a history of blood donation in excess of 500 mL of blood within 30 days prior to Visit 1.
* Have received treatment with an investigational drug or device within 60 days prior to Visit 1.
* Have a positive test for human immunodeficiency virus (HIV) antibodies, Hepatitis B surface antigen or Hepatitis C antibody.
* Are an employee of Omeros, an investigator, a study staff member, or their immediate family member.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Safety | 14 days
  Incidence of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics | Pre-dose and up to 10 days post-dose
  Maximum plasma concentration of OMS643762 following multiple-dose administration
Pharmacokinetics | Pre-dose and up to 10 days post-dose
  Area under the concentration-time curve of OMS643762 following multiple-dose administration
Cognition | Pre-dose and on day 14 of dosing
  Time to complete the Trail Making Test
Cognition | Pre-dose and on day 14 of dosing
  Number of correct responses on the Stroop Color and Word Test
Cognition | Pre-dose and on day 14 of dosing
  Number of correct responses on the Hopkin's Verbal Learning Test-Revised

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yu, MD, Study Director — Omeros Corporation
Locations (1):
- Long Beach, California, United States